CLINICAL TRIAL: NCT01903382
Title: The Association Between Circadian, Weekly, and Seasonal Effects and Time of Surgery on Postoperative Morbidity and Mortality of Patients (Zirkadianest)
Brief Title: Circadian, Weekly and Seasonal Variability of Postoperative Mortality and Morbidity (Zirkadianest)
Status: Completed | Type: Observational
Sponsor: Charite University, Berlin, Germany (Other)
Responsible Party: Principal Investigator, Claudia Spies, Department of Anesthesiology and Intensive Care Medicine CVK/CCM, Charite University, Berlin, Germany, Charite University, Berlin, Germany
Other Study IDs: Zirkadianest
Record Dates: First submitted 2013-07-16; First posted 2013-07-19 (Estimated); Last update posted 2014-11-10 (Estimated); Status verified 2014-11

CONDITIONS: Postoperative Mortality and Morbidity

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Adult patients: All patients undergoing general anesthesia between January 2006 and December 2013

SUMMARY:
Mortality is subject to cyclic variability: circadian, weekly, and seasonal. This has been shown for different populations, different diseases and in different countries, but not for surgical patients. Aim of this study is therefore to investigate the association between circadian, weekly, and seasonal effects time of surgery postoperative mortality of patients undergoing surgery and general anesthesia.

ELIGIBILITY:
Inclusion Criteria:

All Patients who underwent anesthesia within the study time period.

Exclusion Criteria:

none

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: All patients undergoing general anesthesia between January 2006 and December 2013. They are followed up until hospital discharge.
Sampling Method: Non-Probability Sample
Enrollment: 247506 (Actual)
Dates: Start 2006-01; Primary Completion 2014-06 (Actual); Study Completion 2014-06 (Actual)

PRIMARY OUTCOMES:
Postoperative mortality | One year
  The primary objective of this study is to show associations between postoperative mortality and circadian, weekly and seasonal rhythms.
  Electronic patient charts are revised for complete hospital length of stay for time of surgery, co-morbidities, intra-operative data and all-cause in-hospital mortality

SECONDARY OUTCOMES:
Hospital length of stay | One year
  The secondary objective of this is to show associations between hospital length of stay and circadian, weekly and seasonal rhythms. Electronic patient charts are revised for complete hospital length of stay for time of surgery, co-morbidities, intra-operative data and hospital length of stay

CONTACTS AND LOCATIONS:
Overall Officials: Claudia Spies, MD Prof., Study Director — Charite University, Berlin, Germany
Locations (1):
- Department of Anesthesiology and Intensive Care Medicine Campus Charité Mitte and Campus Virchow-Klinikum, Charité - University Medicine, Berlin, State of Berlin, Germany